CLINICAL TRIAL: NCT06297850
Title: Validation of the Accuracy of Continuous Glucose Monitoring Using the Dexcom G7 in Patients With Diabetes in Situations With Circulatory Impairment. A Prospective Observational Study
Brief Title: Accuracy of Continuous Glucose Monitoring in Patients With Diabetes. A Prospective Observational Study
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Rigshospitalet, Denmark (Other); Steno Diabetes Center Copenhagen (Other); Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Casper Pedersen, MD, principal investigator, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: WARD-Glucose Validation v.2.2
Record Dates: First submitted 2024-02-26; First posted 2024-03-07 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus; Dysglycemia; Perioperative Complication; Circulatory; Complications
Keywords: Diabetes Mellitus; Continuous glucose monitoring; Medical devices
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring; Drug Delivery Systems

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Dexcom G7 Continuous Glucose Monitoring (CGM) System (G7) — A CGM device placed on the posterior aspect of the upper arm in which a sensor placed in the skin registers glucose values. Via Bluetooth, these readings are sent to a receiver near the patient every 5 minutes. The CGM system can alert when deviating glucose levels, but will for this observational study be blinding to patients and clinical staff. Thus, the patients' diabetic care will rely on standard practice.
  Other Names: Dexcom G7

SUMMARY:
The goal of this observational study is to investigate the accuracy of the continuous glucose monitoring (CGM) compared to standard point-of-care (POC) blood glucose measurements in patients with diabetes in patients who during their hospital admission can experience circulatory impairment.

The main questions it aims to answer are:

• Do CGM measurements have a decreased accuracy compared to standard blood glucose measurements in periods with circulatory impairment?

Participants will be asked to wear a blinded CGM device (Dexcom G7, Dexcom Inc.) during their stay in the hospital but will receive standard care of their diabetes. The CGM device will be worn for up to 10 days.

DETAILED DESCRIPTION:
This is a prospective observational study on patients living with diabetes who a) undergo surgery at the Department of Vascular Surgery, Rigshospitalet, Denmark and the Surgical Department and Department of Orthopedic Surgery and Traumatology, Bispebjerg and Frederiksberg Hospital, Denmark, or b) are admitted to the intensive care unit (ICU) at Bispebjerg and Frederiksberg Hospital with circulatory impairment.

The study aim is to investigate the accuracy of the Dexcom G7 CGM in patients with diabetes undergoing surgery and in patients at the ICU with circulatory impairment. The glucose readings will be compared to standard practice with POC blood glucose measurements.

Included patients will be asked to wear the CGM device Dexcom G7 for up 10 days.

The study will include 60 patients

This study is part of an overall project that aims to investigate the use of CGM and continuous wireless monitoring of vital signs in patients with diabetes undergoing major surgery. Using this technology, postoperative complications including dysglycaemia can potentially be detected and treated earlier thus improving the perioperative care.

ELIGIBILITY:
Inclusion Criteria:

* Medical history with diabetes mellitus requiring antidiabetic drugs
* Age ≥18 years
* Surgery with estimated surgery time ≥45 minutes with expected stay for at least one night in hospital postoperatively OR
* Admission to the ICU with Circulatory impairment defined as need of vasopressors to maintain a mean arterial pressure (MAP) ≥65 mmHg and peripheral perfusion index <1.5

Exclusion Criteria:

* Local skin symptoms including infection at the posterior aspect of the upper arm that does not allow the sensor to be placed on an unaffected skin area
* Contraindications to skin puncture (arteriovenous fistula for dialysis, post-mastectomy lymphoedema etc)
* Known allergy to plaster used in the CGM device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To the answer of our two research questions, we include both patients with diabetes undergoing surgery, and patients with diabetes admitted to the intensive care unit with circulatory impariment, as described in the criteria above.
  We aim to exclude only patients with direct contraindications to the wear of the CGM.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Agreement between glucose | Perioperatively
  Agreement between glucose readings in mmol/L recorded by the CGM device Dexcom G7 and point-of-care blood glucose measurements (matched pairs within 5 minutes) in the perioperative setting

SECONDARY OUTCOMES:
Agreement between glucose readings when at low glucose levels | Perioperatively
  Agreement between glucose readings in mmol/L recorded by the CGM device Dexcom G7 and point-of-care blood glucose measurements at low glucose levels (<3.9 mmol/l in the POC blood glucose measurement)
Agreement between glucose readings when at normal glucose levels | Perioperatively
  Agreement between glucose readings in mmol/L recorded by the CGM device Dexcom G7 and point-of-care blood glucose measurements at normal glucose levels (>3.9-10.0 mmol/l in the POC blood glucose measurement)
Agreement between glucose readings when at high glucose levels | Perioperatively
  Agreement between glucose readings in mmol/L recorded by the CGM device Dexcom G7 and point-of-care blood glucose measurements at high glucose levels (>10.0 mmol/l in the POC blood glucose measurement)

OTHER OUTCOMES:
Adverse clinical outcomes | 30 days postoperative
  Occurrence and severity of adverse clinical outcomes until 30 days postoperatively according to a set of predefined diagnoses and/or definitions, assessed by physicians at the research unit
Readmission | 6 months postoperatively
  Occurrence of readmission until 6 months postoperatively, assessed by physicians at the research unit
Mortality | 6 months postoperatively
  Occurrence of death until 6 months postoperatively, assessed by physicians at the research unit

CONTACTS AND LOCATIONS:
Overall Officials: Eske K Aasvang, MD, DmSci, Study Director — Dept. of Anaesthesiology, Centre for Cancer and Organ Diseases, Rigshospitalet, Denmark
Locations (4):
- Denmark (4):
  - Department of Anaesthesiology, Centre for Cancer and Organ Diseases, Rigshospitalet, Copenhagen, The Capital Region of Denmark
  - Department of Anaesthesiology and Intensive Care, Bispebjerg Hospital, Copenhagen, The Capital Region of Denmark
  - Department of Orthopaedic Surgery and Traumatology, Bispebjerg and Frederiksberg Hospital, Copenhagen, The Capital Region of Denmark
  - Surgical department, Bispebjerg and Frederiksberg Hospital,, Copenhagen, The Capital Region of Denmark

IPD SHARING:
Plan to Share IPD: No
We do not plan making individual patient data available to researchers outside the study group.